CLINICAL TRIAL: NCT06548126
Title: Evaluation of the Parenting in the Moment Program for Forcibly Displaced Families
Brief Title: Evaluation of the Parenting in the Moment Online Program for Forcibly Displaced Families
Acronym: PIMonline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Abigail Gewirtz, Co-Director of REACH and Professor, Psychology, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90FA3009
Record Dates: First submitted 2024-05-02; First posted 2024-08-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Child Safety; Coercion; Child Wellbeing; Adjustment; Parenting; Post Traumatic Stress Disorder; Mental Health; Child Maltreatment; Trauma; Emotional Regulation
Keywords: Forced displacement; Refugees; Parenting Program; Immigrant Parenting Program; Refugee Parenting Program
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Psychological Well-Being; Wounds and Injuries; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Families will be recruited using stratified random sampling within the four PIM language groups; 180 families will be recruited from each (English, Spanish, French, Arabic), from which 90 families will be assigned to the intervention. This study will randomly select intervention and control families as they enter the study following a 1:1 randomization scheme.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Study Staff members involved with contacting families for scheduling purposes, administering the Family Interaction Tasks and administering Target Child surveys are prevented from having knowledge of individual participants' randomization assignment. The principle investigator and outcome assessor are also masked and prevented from having knowledge of individual participants' randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting Intervention (Experimental): Participants will receive the PIMonline program and a list of Parenting resources.
  Interventions: Behavioral: Online Parenting Program
- Control (Placebo Comparator): Participants will receive a list of Parenting resources. Once the study period ends, they will be given access to the PIMonline program.
  Interventions: Other: No online parenting program

INTERVENTIONS:
Behavioral: Online Parenting Program — Online Parenting Program comprised of 12 online modules. Caregivers do one module per week for 12-15 weeks; each unit takes about 20 minutes to do. The Caregiver also practices the tools they learn for Parenting their Children between sessions.
  Other Names: PIMonline; PIM Treatment; Parenting in the Moment
  Arms: Parenting Intervention
Other: No online parenting program — List of Parenting resources.
  Other Names: Control; Placebo
  Arms: Control

SUMMARY:
This Randomized Controlled Trial will test the effectiveness of the Parenting in the Moment (PIM) online parenting program for parents with experiences of forced displacement.

The primary objective of this study is to conduct a summative (impact) evaluation of the PIM online parenting program as an in-home parent, skill-based program for parents of school-aged children, using a randomized controlled trial research design with community partnerships that inform the research throughout. The longer-term objectives are to build the evidence-base for in-home parent skill-based programs with strong empirical support (i.e., eligible for listing on the Families First Clearinghouse) and increase access to parenting programs for forcibly displaced families thereby improving child safety and wellbeing and strengthening their public health support.

720 families will be recruited with forced migration backgrounds and within 10 years of arrival in the USA; 360 families will be assigned to the PIMonline program and 360 to a family resource list only, wait-list control group. Families will be recruited using stratified random sampling within the four PIM language groups: English, Spanish, Arabic, French. Within each language, half the families will be assigned to the PIMonline intervention program and the other half will be assigned to receiving a Family Resource List with access to the PIMonline program once the study ends.

One parent and one child per eligible family may participate. Data collection with participating families will take place at baseline (T1), 4-months after baseline (T2) and finally, 16 months after baseline (T3). Data collection includes caregiver online surveys, caregiver and child Zoom recorded Family Interaction Task conversations and interviewer administered child surveys for children aged 8-12 at each time point. Standardized, reliable and valid measures in the four languages will be used to assess change in outcomes through the surveys. Longitudinal growth curve analysis will be used to test PIM intervention effects. Our extensive dissemination plan involves nationwide community partners in child welfare and services to forcibly displaced families.

DETAILED DESCRIPTION:
Families may contact Study Personnel with any questions at any time. All elements of this study are completed online or virtually (over phone/zoom conference).

Recruitment efforts will be purposive and snowballing. Recruitment efforts will take place through social media and word of mouth campaigns. Communities will be reached out to broadly via word-of-mouth (with electronic and printed flyers) through the help of Community Advisory Board members, community partners and other groups and organizations that provide direct interaction and services to immigrant and refugee populations in the US. The project will also be advertised on the REACH Institute website at Arizona State University. In addition to flyers, video ads will also be used on social media platforms.

Interested Caregivers will complete an online eligibility screening form to verify eligibility according to the specified criteria. Caregivers who are ineligible will be thanked for their interest and provided with a Family Resource List. If Caregivers meet criteria for inclusion on the screening form, their information will be verified for authenticity. In order to avoid enrollment of robots or false positive cases, quality control measures will be carried out. These include checking IP address; the use of hidden questions that robots will respond to in efforts of identifying robots (real humans cannot see these hidden questions but robots can); validity questions (e.g. child gender; child DOB, caregiver relationship) for cross-comparing and checking validity of the data/respondent in addition to an open text box (asking country of origin). Any received forms suspected of being robots, or possibly invalid, will have a Study Staff member contact the family to verify authenticity of enrollment by reviewing some information provided in the eligibility screening form to ensure it is authentic input and not false or fabricated.

Caregivers who are eligible and verified to be real will then receive a study welcome email with further information about the project and a link to a personalized consent form to sign electronically. Upon signing the electronic consent form, families will automatically move to the pretest survey. The pretest survey asks a variety of questions that include: demographics, Parenting, adjustment, family values, attitude, trauma-related questions, spirituality, self-report of Parenting, self-report of mental health and well-being, and Caregiver reporting on Child mental and behavioral health problems.

After the Caregiver Pretest survey is submitted, a Study Staff member will contact the family to schedule Zoom recorded Family Interaction Task conversations between the Caregiver and Target Child, and (for children aged 8-12) the Target Child's survey, which will be administered by Study Team Staff. Child Assent will be recorded along with verifying Parent Permission for the Child to participate when the family is called for their scheduled Family Interaction Task conversation and Target Child survey.

The Family Interaction Task conversation activities ask the Caregiver and Target Child to have two conversations: 1) about problem solving (problems that may be stressful for Parents and kids) and 2) about the migration experience (things the Child might be experiencing following migrating to the US).

The Target Child survey asks the Child questions related to the Child's mental and behavioral health as well as some trauma-related questions.

After all pretest data collection (Baseline Caregiver survey, Family Interaction Tasks and Target Child survey) is completed, the Caregiver is randomized to either a) the intervention condition or b) the waitlist control condition.

Caregivers assigned to the intervention condition will receive a welcome email with a Family Resource List and instructions on how to start the Parenting in the Moment online program.

Caregivers assigned to the waitlist control condition will receive an email with a Family Resource List.

Caregiver surveys, Family Interaction Tasks and Child surveys take place at times: 0- baseline, 4 months-posttest and 16 months posttest.

After intervention families complete the PIMonline Parenting program, they will provide Course Feedback and receive a Certificate of Completion.

After the study period ends, the waitlist control group will be emailed instructions on how to access the PIMonline program.

Study instrument codebooks (for each survey and the coding of Family Interaction Tasks) detailing descriptions of each variable used, including the source of the variable, coding information, and ranges (if relevant) will be saved and stored for reference.

Primary objectives will be analyzed using linear growth curves with three waves of survey scores.

Descriptive statistics, ANOVA, and crosstabs to examine the reach of social media and other recruitment strategies will be used. And descriptive statistics will be used to report participation and satisfaction.

To manage data, a secure website and server maintaining stringent HIPAA-compliant levels of encryption and data storage, and sophisticated data management and collection features will be employed. The data manager will regularly download data from Redcap to check for errors, duplicates, and missing information. Data will be cleaned, scored, and stored in SPSS or Excel formats. Confidentiality is addressed by removing personal identifiers from database files and restricting access authorization to a specific set of project personnel only. Databases generated for analysis will be de-identified prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

1. The person is a primary Caregiver to a Child age 6 - 12 years in their care and living with them at least half the time
2. The Caregiver is at least 18 years of age
3. The Caregiver is able to do a program delivered in English, Spanish, Arabic or French, and to answer questions in English, Spanish, Arabic or French.
4. The Caregiver resides in the United States
5. The Caregiver has reliable access to a smart phone, tablet, or computer with stable internet access.
6. One Parent, not necessarily the PCG, has experienced forced displacement in the past 10 years
7. The Parent is able to consent for self and Child If the PCG does not have the legal right to provide Parent permission for the Child to participate, the Child's legal Parent/Caregiver can provide consent while the PCG actively participates in the study with the Child.
8. The Child is able to answer questions in English, Spanish, Arabic or French.

Exclusion Criteria:

1. Prisoners
2. Impaired decision-making capacity
3. Disclosed active psychosis of Parent or Child
4. Open Child protection case for abuse or neglect in the family

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Child Safety | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: Child Abuse Screening Tool (ICAST-T attitudes to punishment scale)
Child Safety | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: UNICEF (Multiple Indicator Cluster Survey (MIC5)
Child Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: Parent report on child - Eyberg Child Behavior Inventory (ECBI)
Child Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: Parent report on child - Revised Child Anxiety and Depression Scale (RCADS).
Child Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  For child wellbeing this is what it reads: Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: Child report on self- Revised Child Anxiety and Depression Scale (RCADS).
Child Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  For child wellbeing this is what it reads: Structural equation modeling (SEM) growth curve analyses on child outcomes will be employed. The following evidence-based measures will be used to measure change and determine child safety outcomes as a result of the intervention: Child report on self- UCLA Child Trauma plus PTSD.
Adult Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: Parent Locus of Control (PLOC-SFR).
Adult Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: Patient Health Questionnaire (HTQ, Diagnostic and Statistical Manual-5) PTSD Events.
Adult Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: World Health Organization (WHO5).
Adult Wellbeing | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: Harvard Trauma Questionnaire (HTQ-5) Trauma Events.
Covariates and control variables | 0-Baseline (timepoint 1)
  Demographics measure to include: gender, age, racial and ethnic identity of caregivers and children; language(s) spoken; education, employment, income, and information about the migration experience, including countries of origin, reasons for fleeing.
Caregiver Satisfaction with the intervention | 4-month Posttest (timepoint 2)
  Descriptive statistics and a Parenting in the Moment acceptability and feasibility survey.
Emotion Coaching | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Observational Coder ratings will yield reliable and valid measures of parenting practices with short- and long-term predictive validity for child and parent outcomes. Rating will yield the primary construct: emotion socialization. Scale scores yield reliable Cronbach alphas (ranging from .74-.92) and interrater reliabilities in the 70-80% range.
Problem Solving | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Observational Coder ratings will yield reliable and valid measures of parenting practices with short- and long-term predictive validity for child and parent outcomes. Rating will yield the primary construct: positive parenting (family problem-solving, skill encouragement, positive involvement, monitoring). Scale scores yield reliable Cronbach alphas (ranging from .74-.92) and interrater reliabilities in the 70-80% range.

SECONDARY OUTCOMES:
Adult Wellbeing secondary outcomes | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: Difficulties in Emotion Regulation Scale (DERS).
Adult Wellbeing secondary outcomes | 0-Baseline (timepoint 1); 4-month Posttest (timepoint 2); 16-month Posttest (timepoint 3)
  Structural equation modeling (SEM) growth curve analyses on Caregiver outcomes will be employed. The following evidence-based measures will be used to measure change and determine adult wellbeing outcomes as a result of the intervention: Coping with Negative Emotions Scale (CCNES).

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gewirtz, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No